CLINICAL TRIAL: NCT07397598
Title: Peer Support to Enhance Care for Liver Transplant Recipients Who Had Alcohol-Associated Liver Disease
Brief Title: Peer Support for Liver Transplant Recipients With History of ALD
Acronym: THRIVES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00466249; P50AA027054 (NIH)
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Alcohol Use Disorder; Alcohol Related Liver Disease; Liver Transplant Recipient
Keywords: Alcohol use disorder; Alcohol Related Liver Disease; Liver transplant recipient; Peer support specialist
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer Support Specialist (PSS) (Experimental)
  Interventions: Behavioral: Peer Support

INTERVENTIONS:
Behavioral: Peer Support — The study will recruit PSS based on lived experiences with ALD/LT and interpersonal skills. The PSS will receive tailored skills training from the study team in areas such as delivering brief counseling, active listening, and maintaining confidentiality.
  Participants will meet regularly with a PSS between standard clinic visits throughout a one-year study period. The PSS will deliver brief counseling interventions at each session. Study investigators will meet with the PSS at scheduled intervals to review progress. Study investigators will also review up to 20% of the audio recordings of sessions between PSS and study participants to assess fidelity to the intervention protocol.

SUMMARY:
Liver transplant (LT) recipients with a history of alcohol-related liver disease (ALD) may encounter various psychosocial and medical challenges during post-LT recovery, even beyond the initial post-transplant period. Effective and sustainable interventions will be crucial for improving patient outcomes. This clinical trial will examine the impact of peer support specialists (PSS) on the recovery experience of individuals who received LT for ALD. The trial seeks to answer two main questions:

* Are LT recipients who work with PSS less likely to resume alcohol use or tend to drink less overall?
* Do LT recipients who work with PSS engage more with recommended medical care and have better overall survival?

DETAILED DESCRIPTION:
In the United States, ALD is the most common indication for LT. Resuming alcohol use is a major concern for all LT recipients with a history of ALD, with estimates ranging from 16% to 49% and increasing with more time since LT. Although most LT programs have required pre-LT alcohol treatment, post-LT services have been far more heterogeneous, despite the potentially severe consequences of alcohol relapse during this period. The present study proposes implementing and evaluating a care model for LT recipients with a history of ALD after the first post-LT year. The investigators will conduct a single-arm clinical trial to integrate PSS into routine medical care starting in years 2 through 4 following LT. The study will recruit PSS based on lived experiences with ALD/LT and interpersonal skills. The PSS will first receive tailored skills training from the study team in areas such as delivering brief counseling, active listening, and maintaining confidentiality. The PSS will then meet with study participants at regular intervals between standard clinic visits. The investigators will follow participants working with PSS for 1 year and compare the participants with a historical control group of transplant recipients without PSS to determine whether the intervention improves outcomes. Key endpoints will include alcohol use (by self-report and biomarker), retention in post-transplant medical care, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* English speakers
* Received a liver transplant for alcohol-associated liver disease
* Has 1 to 3 years of continuous alcohol abstinence at the time of trial entry

Exclusion Criteria:

* Liver transplant recipients without a history of alcohol-associated liver disease
* Inability to provide informed consent
* Active participation in a separate intervention trial for alcohol use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Alcohol Consumption | Up to 1 year
  Any use or excessive use (i.e., >7/>14 drinks per week for women/men) by biomarker or self-report

SECONDARY OUTCOMES:
Liver Transplant Medical Treatment Engagement | Up to 1 year
  Proportion of kept/scheduled LT follow-up medical appointments
Overall Post-Liver Transplant Survival | Up to 1 year
  All-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Po-Hung Chen, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient reported outcomes and phosphatidylethanol biomarker results
Time Frame: Data will be shared with the general research community at the time of an associated publication, or the end of the award/grant period, whichever comes first. Data will be shared indefinitely.
Access Criteria: Summaries of NIAAA Data Archive (NIAAADA) data are publicly available to anyone through the NDA Query Tool without an account. Access to individual participant data and supporting documentation is limited to qualified researchers who create an NDA account and submit a Data Access Request (DAR), including completion of the NDA Data Use Certification (DUC). Requests are reviewed by a NIAAA committee to ensure responsible data use. Individual-level data are accessed through the NDA Query Tool once approval is granted.
URL: https://www.niaaa.nih.gov/research/data-archive-and-resources/niaaa-data-archive